CLINICAL TRIAL: NCT05549765
Title: The Effectiveness and Safety of Pharmacopuncture on Inpatients With Tension Headache Caused by Traffic Accidents: A Pragmatic Randomized Controlled Trial
Brief Title: The Effectiveness of Pharmacopuncture on Acute Tension Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2022-11
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Tension Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacopucture on suboccipital muscles (Experimental): The Pharmacopucture group will recieve 3 sessions of Pharmacopucture on suboccipital muscles; on second, third, fourth day after hospitalization. A trained doctor of Korean medicine with at least 3 years of clinical experience are going to conduct the pharmacopucture.
  The Pharmacopucture group will also be treated with other Korean medical treatment everyday: acupuncture, chuna and Korean herbal medicine.
  Interventions: Procedure: Pharmacopuncture; Procedure: Korean medical treatment
- Korean medical treatment (Active Comparator): The control group will be received Korean medical treatment everyday after hospitalization: acupuncture(except on suboccipital parts), chuna, pharmacoacupuncture and Korean herbal medicine
  Interventions: Procedure: Korean medical treatment

INTERVENTIONS:
Procedure: Pharmacopuncture — Pharmacopuncture is a treatment that combines 2 of the most frequented Korean medicine treatment methods - traditional acupuncture and herbal medicine - by injecting herbal medicine extract at acupoints.
  Arms: Pharmacopucture on suboccipital muscles
Procedure: Korean medical treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine

SUMMARY:
This study is a double blind, randomized controlled trail. condition/disease: acute tension headache treatment/intervention: Pharmacopuncture

DETAILED DESCRIPTION:
"Pharmacopuncture is a treatment that combines 2 of the most frequented Korean medicine treatment methods - traditional acupuncture and herbal medicine - by injecting herbal medicine extract at acupoints.

This treatment is known to be an important part of Korean medicine treatment. However, there has been no specific value for the effect of this treatment.

Therefore, the investigators are going to conduct a randomized controlled trials to verify the efficacy and safety of Pharmacopuncture. From September 2022 to December 2023, the investigators are going to collect 80 inpatients who are suffering from Tension headache with the numeric rating scale(NRS) over 5 after injury by acute traffic accident(TA). For experimental group(n=40), the investigators will conduct Pharamacopuncture on suboccpital muscle three times(on 2nd, 3rd and 4th day of hospitalization) and other Korean medical treatment. For control group(n=40), just Korean medical treatment except Pharamacopuncture on suboccpital muscles will be conducted.

For these two groups, the investigators will compare Numeric Rating Scale(NRS) of headache, NRS of Neck pain, Headache Disability Index(HDI), Headache Impact Test-6(HIT-6), EuroQol 5-Dimension (EQ-5D-5L) and Patient Global Impression of Change (PGIC)."

ELIGIBILITY:
Inclusion Criteria:

* Patients who needs hospitalization due to acute tension headache that occurred within 7 days after traffic accident
* Patients with NRS ≥ 5 for headache
* Patients aged 19-69 years on the date they sign the consent form
* Patients who provide consent to participate in the trial and return the informed consent form

Exclusion Criteria:

* Patients with a specific serious disease that may cause headache: malignancy, cerebral hemorrhage, dural hematoma, etc.
* Patients with progressive neurological deficits or with severe neurological symptoms- Patients who have had surgery or procedures within the last three weeks
* The cause of pain is due to soft tissue disease, not the nerve system disease: trigeminal neuralgia, glossopharyngeal neuralgia, etc.
* Patients with other chronic conditions that may interfere with the interpretation of the therapeutic effects or results: cardiovascular disease, kidney disease, diabetic neuropathy, dementia, epilepsy, etc.
* Patients who are taking steroids, immunosuppressants, mental illness drugs, or other drugs that may affect the results of the study
* If pharmacopuncture and acupuncture is inadequate or unsafe: patients with hemorrhagic, receiving anticoagulants, severe diabetes and cardiovascular disease
* Patients who are pregnant or planning to become pregnant
* Patients with a serious mental illness
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement
* Other patients whose participation in the trial is judged by a researcher to be problematic

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of headache | Change from baseline NRS at 4 days
  The extent of headache and discomfort will be assessed by using NRS. NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their headache and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Numeric Rating Scale(NRS) of Neck pain | Baseline(day2), day3, day4, day of discharge(up to 14days), week 8
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their leg pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Headache Disability Index(HDI) | Baseline(day2), day4, day of discharge(up to 14days), week 8
  The HDI is a 25-item, self-report headache disability measure that has good internal consistency reliability and strong long-term test-retest stability.
Headache Impact Test-6(HIT-6) | Baseline(day2), day4, day of discharge(up to 14days), week 8
  The HIT-6 items measure the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning and psychological distress. The HIT-6 also measures the severity of headache pain.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Baseline(day2), day4, day of discharge(up to 14days), week 8
  The EQ-5D is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, the investigators will use the Korean version of the EQ-5D, which has been demonstrated to be valid.
Patient Global Impression of Change(PGIC) | day4, day of discharge(up to 14days), week 8
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, phD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No